CLINICAL TRIAL: NCT01661647
Title: (Étude de la cinématique Tridimensionnelle du Genou Humain Lors de Gestes Sportifs et de la Vie Courante)
Brief Title: 3D Kinematic Assessment of the Human Knee During Physical and Daily Life Activities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Eiffel Medtech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 12.005
Record Dates: First submitted 2012-07-16; First posted 2012-08-09 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: 3D Knee Kinematics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D knee kinematic assessment (Experimental): 3D knee kinematic assessment under local anesthesia
  Interventions: Device: 3D knee kinematic assessment under local anesthesia

INTERVENTIONS:
Device: 3D knee kinematic assessment under local anesthesia — 3D knee kinematic assessment under local anesthesia

SUMMARY:
Problem : Precise and personalized 3D knee kinematic assessment during physical and daily life activities is a challenge; therefore, it was never performed on an important number of individuals. However, a better understanding of 3D knee kinematics during such activities would allow a better understanding of this often injured joint.

Hypothesis: A new system using personalized 3D bone imaging and a percutaneous bone fixation device that can be used under local anesthesiaallows for precise and reproducible assessment of 3D knee kinematics during physical and daily life activities.

Objectives :

* To study human knee 3D kinematics during dynamic activities using a novel minimally invasive measuring system
* Investigate the correlations between standard clinical knee laxity tests and measured 3D knee kinematics during dynamic activities

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting knee arthroscopy under local anesthesia for a medial meniscal tear

Exclusion Criteria:

* Active infection
* Severe swelling of the knee
* Knee flexion contracture
* Knee flexion less than 120 degrees
* Gross limping
* Inability to perform the various motor tasks required by the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
3D knee kinematics | On the day of the surgery, before knee arthroscopy
  The investigators will investigate if 3D knee kinematics can be precisely and safely measured under local anesthesia during various motor tasks (walking, squatting, pivoting, jumping): kinematic data will be analyzed in search of signs of artefact movement and kinematic aberrations, which would indicate problems with the measurement system.

SECONDARY OUTCOMES:
Correlation of kinematic data with clinical laxity tests | On the day of surgery, before knee arthroscopy
  With the kinematic measurement device attached to the bones of the lower limbs, various knee laxity tests will be performed by a physician while the kinematics of the knee are recorded; correlations will be sought between the subjective evaluation of the physician and the kinematic data.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lavoie, MD MSc FRCSC, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada